CLINICAL TRIAL: NCT01192230
Title: A Phase 2 Study of Gefitinib Compared With Pemetrexed/Cisplatin in Advanced Non-Small Cell Lung Cancer Patients
Brief Title: Study of Endostatin Combined With Docetaxel in the Treatment of Advanced Non-small Cell Lung Cancer Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Base for drug clinical trials, Fudan University Cancer Hospital, Department of Medical Oncology,Fudan University Cancer Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EndoDocNSCLC
Record Dates: First submitted 2010-08-04; First posted 2010-09-01 (Estimated); Last update posted 2010-09-16 (Estimated); Status verified 2010-08

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Objective response rate; Disease control rate; Disease free survival; Overall survival; Quality of Live; Nonsmall cell lung cancer; toxicity
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Endostatins; Docetaxel

INTERVENTIONS:
Drug: Endostatins — 7.5mg/m2 qd *14d,q3w
Drug: Docetaxel — 75mg/m2 D1, q3w,4-6cycles

SUMMARY:
The purpose of this study is to examine the efficacy and safety of endostatin combined with Docetaxel in advanced Non-Small-Cell Lung Carcinoma (NSCLC) patients failure to first-line or second-line chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were diagnosed by the histologic, cytologic diagnosis of IIIB (malignant hydrothorax or hydropericardium) or IV non-small cell lung cancer
* ≥ 18 years old
* patients who have received more than one regimen of platinum-based chemotherapy; patients who have received EGFR monoclonal treatment could also be enrolled
* At least one target lesion diameter spiral CT ≥ 1 cm, or the common CT ≥ 2 cm, and can be measured by imaging tools
* have an interval of more than 4 weeks from the last chemo- or radio-therapy; 2 weeks from the last targeted therapy
* ECOG 0-2
* Expected life time longer than 3 months
* Normal laboratory values:

  * leucocyte≥ 4×109/L
  * neutrophil≥ 1.5×109/L
  * platelet≥90×109/L
  * Hemoglobin≥ 9g/L
  * ALT and AST ≤3×ULN (≤5×ULN if liver metastasis)
  * serum creatinine<1.5 mg/dl
  * bilirubin <1.5×ULN
* No allergy to biological drug
* Sign the consent forms

Exclusion Criteria:

* Patients who have previously received Docetaxel or anti-VEGF inhibitors
* Severe symptomatic heart disease
* Female patients during their pregnant and lactation period, or patients without contraception
* Severe uncontrolled infection
* Uncontrolled neurologic or psychiatric disease; Uncontrolled primary or metastatic brain tumor
* Patients with other malignant tumor,except for basal cell carcinoma,squamous cell carcinoma and carcinoma in situ
* Patients have accepted other clinical trials

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2009-06; Primary Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Response rate | six weeks
Progression free survival | six weeks
Overall survival | three months

SECONDARY OUTCOMES:
Quality of Life | six weeks
  EORTC QLQ-C30(v3.0)

CONTACTS AND LOCATIONS:
Overall Officials: Jianhua Chang, MD,PhD, Principal Investigator — Fudan University affiliated cancer hospital
Locations (1):
- Cancer hospital Fudan University, Shanghai, Shanghai Municipality, China